CLINICAL TRIAL: NCT01060904
Title: A Phase 1 Dose-Escalation Safety Study of Brentuximab Vedotin in Combination With Multi-Agent Chemotherapy as Frontline Therapy in Patients With Hodgkin Lymphoma
Brief Title: A Phase 1 Study of Brentuximab Vedotin Combined With Multi-Agent Chemotherapy for Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-009
Expanded Access: NCT01196208 (No longer available)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Disease, Hodgkin
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Disease, Hodgkin; Hematologic Diseases; Immunotherapy; Lymphoma; monomethyl auristatin E
MeSH Terms: conditions — Hodgkin Disease; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): brentuximab vedotin combined with ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine)
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin; Drug: vinblastine; Drug: dacarbazine; Drug: bleomycin
- 2 (Experimental): brentuximab vedotin combined with AVD (doxorubicin, vinblastine, dacarbazine)
  Interventions: Drug: doxorubicin; Drug: vinblastine; Drug: dacarbazine; Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 0.6-1.2 mg/kg IV every 2 weeks
  Other Names: SGN-35
  Arms: 1
Drug: doxorubicin — 25 mg/m2 IV every 2 weeks
Drug: vinblastine — 6 mg/m2 IV every 2 weeks
Drug: dacarbazine — 375 mg/m2 IV every 2 weeks
Drug: bleomycin — 10 units/m2 IV every 2 weeks
  Arms: 1
Drug: brentuximab vedotin — 0.9-1.2 mg/kg IV every 2 weeks
  Other Names: SGN-35
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety profile of brentuximab vedotin in combination with multi-agent chemotherapy in treatment-naive Stage IIa or IIb-IV Hodgkin lymphoma. It is a phase 1, two-arm, open-label dose escalation study designed to define the maximum tolerated dose, pharmacokinetics, immunogenicity and anti-tumor activity of brentuximab vedotin in combination with frontline therapy.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive Hodgkin lymphoma, Stage IIa or IIb-IV
* Measurable disease of at least 1.5 cm
* Eastern Cooperative Oncology Group performance status <3

Exclusion Criteria:

* History of another primary malignancy that has not been in remission for at least 3 years
* Known cerebral/meningeal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | Through 1 month after last dose

SECONDARY OUTCOMES:
Brentuximab vedotin concentration in blood | Through 1 month after last dose
Antitherapeutic antibodies in blood | Through 1 month after last dose
Best clinical response | Through 1 month after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hunder, MD, Study Director — Seagen Inc.
Locations (4):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
- British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Younes A, Connors JM, Park SI, Fanale M, O'Meara MM, Hunder NN, Huebner D, Ansell SM. Brentuximab vedotin combined with ABVD or AVD for patients with newly diagnosed Hodgkin's lymphoma: a phase 1, open-label, dose-escalation study. Lancet Oncol. 2013 Dec;14(13):1348-56. doi: 10.1016/S1470-2045(13)70501-1. Epub 2013 Nov 15. PMID 24239220